CLINICAL TRIAL: NCT07267286
Title: Efficacy of Tirellizumab Combined With TP Neoadjuvant Therapy in the Treatment of Early Oral Squamous Cell Carcinoma (cT1-2N0M0) Versus Standard Therapy: a Randomized Controlled, Single-center Exploratory Clinical Study
Brief Title: Tirellizumab Combined With TP Neoadjuvant Therapy in the Treatment of Early Oral Squamous Cell Carcinoma （HNC-SYSU-005）
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-1018-01
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2024-12

CONDITIONS: HNSCC; PD-1
Keywords: HNSCC; PD-1
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirellizumab combined with TP neoadjuvant therapy combined with surgery (Experimental): All subjects in the experimental group were given 200mg of tirellizumab before surgery, intravenous infusion on the first day of each cycle, 1 cycle every 3 weeks (Q3W), a total of 2 cycles, in which the operation was scheduled for 29-56 days after the first administration; At the same time, the administration cycle of carboplatin and albumin-bound paclitaxel was 1 cycle every 3 weeks (Q3W). Carboplatin was administered on the first day of each cycle, 300mg/m2, intravenous infusion, infusion time ≥1h; Albumin-bound paclitaxel 260mg/m2 was administered on the first day of each cycle for 30min intravenously.
  Interventions: Drug: Tirellizumab combined with carboplatin and albumin-paclitaxel neoadjuvant therapy+surgery
- Traditional surgery (Active Comparator): The control group was treated according to NCCN guidelines, including radical resection of oral cancer combined with selective neck lymphatic dissection.
  Interventions: Procedure: Traditional surgery

INTERVENTIONS:
Drug: Tirellizumab combined with carboplatin and albumin-paclitaxel neoadjuvant therapy+surgery — Tirellizumab 200mg will be administered on day 1 of each 21-day cycle (once every 3 weeks). Tirelizumab will be administered by intravenous infusion using an intravenous catheter containing a sterile, pyrogen free, low protein-binding, 0.2 or 0.22 micron diameter embedded filter or auxiliary filter.
  As a routine precaution, patients must be monitored for at least 60 minutes in an area equipped with resuscitation equipment and first aid medication after the infusion of tirellizumab during cycle 1 and day 1 of cycle 2. Starting with cycle 3, it is required to be monitored for more than 30 minutes (inclusive) in an area equipped with resuscitation equipment and first aid medication.
  The first infusion (day 1 of Cycle 1) will be completed within 60 minutes; If it is well tolerated, subsequent infusions can be completed within 30 minutes, which is the minimum time allowed by the infusion. Tirellizumab should not be administered at the same time as any other drug.The surgical method was exte
  Arms: Tirellizumab combined with TP neoadjuvant therapy combined with surgery
Procedure: Traditional surgery — The control group was treated according to NCCN guidelines, including radical resection of oral cancer combined with selective neck lymphatic dissection
  Arms: Traditional surgery

SUMMARY:
Efficacy of Tirellizumab combined with TP neoadjuvant in the treatment of early Oral squamous cell carcinoma (cT1-2N0M0) versus standard treatment: a randomized controlled, single-center exploratory clinical study. Surgery is usually the preferred treatment for early oral squamous cell carcinoma (OSCC). However, the five-year survival rate of early oral cancer is only 75.8%, which is still not satisfactory compared with breast cancer and lung cancer. It is an urgent problem to explore the treatment mode of early oral squamous cell carcinoma patients. This study intends to conduct neoadjuvant therapy of tirellizumab, carboplatin and albumin-bound paclitaxel (TP) in patients with cT1-2N0M0 oral squamous cell carcinoma after neoadjuvant immunotherapy and standard surgical treatment (radical resection of oral cancer + selective neck lymph dissection). A randomized controlled, single-center exploratory clinical study compared with traditional radical resection of oral cancer plus selective neck lymph dissection was conducted to investigate its effectiveness through the difference of 2-year event-free survival (EFS).

This study plans to include 60 patients with early oral squamous cell carcinoma. The subjects will press 1: The proportion of 1 was randomly divided into Tirellizumab combined with TP neoadjuvant therapy combined with surgery (experimental group) and traditional surgery (control group). Tumor tissues, adjacent tissues, whole blood samples, saliva samples and stool samples of patients were collected to observe the imaging and pathological changes before and after treatment. Meanwhile, clinical information of patients was collected. Such as postoperative function and other quality of life indicators, pathological grade, stage, treatment, prognosis, serology, imaging, etc., the main evaluation and comparison of the experimental group and the control group of 2-year event-free survival (EFS) and 5-year overall survival (OS).

DETAILED DESCRIPTION:
oral squamous cell carcinoma (OSCC) is one of the most common cancers in the world, with about 900,000 new cases and 500,000 deaths in 2020, of which about 30-40% are early stage cancers [1, 2]. According to the 2024 NCCN guidelines and 2023 CSCO guidelines, surgery is the main treatment for early oral cancer, and patients with high-risk factors receive adjuvant radiotherapy and chemotherapy after surgery. It has been reported in literature that the 5-year OS of early stage (T1-2N0M0) OSCC is 75.8% [3], among which the 5-year OS of T2N0 OSCC patients is only 72%. The 2-year DFS is only 72%[4]. Clinical studies have shown that the 5-year survival rate of stage I and II in breast cancer patients is 99.2% and 93.1% respectively, while the 5-year survival rate of early lung cancer can reach more than 92% [5]. In comparison, the 5-year survival rate of early oral cancer (cT1-T2) is greatly reduced. Therefore, it is necessary to explore new therapeutic modalities to improve the prognosis of cT1-2N0M0 oral cancer.

With the rise of immunotherapy, patients with advanced head and neck squamous cell cancer are also benefiting. Antibodies to PD-1 or PD-L1 have demonstrated clear anti-tumor activity and safety in multiple cancer types, including melanoma, lung cancer, and head and neck cancer [6, 7]. In both first-line and second-line therapies for oral cancer, Nivolumab (PD-1 inhibitor) and Pembrolizumab (PD-1 inhibitor) have achieved good clinical efficacy, with response rates of 13.3% and 16.4% in Phase II clinical studies, respectively [7,8]. Multiple studies have shown that compared with advanced tumors, early tumors have smaller tumor load and heterogeneity, lower systemic immunosuppression, and more tumor-related T cell infiltration, and PD-1 inhibitors can achieve a higher response rate in neoadjuvant therapy for early solid tumors than for advanced tumors [9-11]. Although there is a lack of research on immunotherapy for early oral cancer, PD-1 inhibitors show good effects in early lung cancer and early triple-negative breast cancer, and EFS is significantly improved [12,13].

Data from our study showed that in 104 patients who received preoperative PD1 monoclonal antibody combined with chemotherapy neoadjuvant therapy, the postoperative pathological complete response (pCR) rate was 47.1%, and the major pathological response (MPR) rate was 65.4% (Figure 1). The 2-year estimated DFS rates were 89.7% and 75.51%, respectively, in the neoadjuvant and conventional surgical treatment cohort, while the 2-year estimated OS rates were 94.5% and 81.2%, respectively (Figure 2).

Figure 1 Postoperative pathological remission of the neoadjuvant exemption cohort FIG. 2 Prognosis of neoadjuvant immunity cohort compared with conventional surgery

Tirellizumab is a humanized IgG4 monoclonal antibody against PD-1, which has high affinity and binding specificity for PD-1. Its modification of Fc segment reduces the antigen-clearing effect of macrophages induced by mediated immune cell crosslinking, and enhances anti-tumor activity. The efficacy of Tirelizumab against tumors has been proven in the treatment of a variety of solid tumors, and its Disease control rate (DCR) can reach 50-80%[14,15]. As a uniquely modified PD-1 inhibitor, Tirellizumab may be safer and more effective in oral cancer. Paclitaxel combined with carboplatin is the first-line protocol for the treatment of recurrent or metastatic oral and oropharyngeal squamous cell carcinoma, and the induction chemotherapy of carboplatin combined with paclitaxel can provide complete and partial response rates of 8% to 33% and 50% to 85%, respectively [16]. Combination immunotherapy, especially immunochemotherapy, has shown better response rate in a variety of cancers, so Tirellizumab combined with carboplatin and paclitaxel has a strong application in oral cancer [7,8,16].

Based on the above research background, we believe that PD-1 (Tirellizumab) combined with carboplatin and albumin-bound paclitaxel has a good application prospect in resectable head and neck squamous cell carcinoma. Therefore, we designed this controlled study to explore the efficacy and safety of PD-1 (tirellizumab) combined with carboplatin and albumin-bound paclitaxel in patients with early oral squamous cell carcinoma before surgery, and to provide a new way to further improve the prognosis of patients with resectable head and neck squamous cell carcinoma. To provide valuable information for planning prospective clinical trials of anti-PD-1 and other immunotherapies combined with chemotherapy in perioperative and advanced disease Settings in patients with oral squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early oral squamous cell carcinoma diagnosed as T1-2N0M0 according to the eighth edition of AJCC TNM stage;
* No history of other malignant tumors;
* 18-75 years old;
* Baseline inspection is normal:

  1. The absolute value of neutrophil (ANC) ≥1.5x109/L in the past 14 days without the use of granulocyte colony-stimulating factor;
  2. Platelets ≥100×109/L without blood transfusion in the past 14 days;
  3. Hemoglobin >9g/dL in the last 14 days without blood transfusion or use of erythropoietin;
  4. Total bilirubin ≤1.5× upper limit of normal (ULN);
  5. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) in ≤2.5×ULN (patients with liver metastases allowed ALT or AST ≤5×ULN);
  6. Serum creatinine ≤1.5×ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥60 ml/min;
  7. Good coagulation function, defined as International standardized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN;
  8. Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. If baseline TSH is outside the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled;
  9. The myocardial enzyme profile is within the normal range (if the researchers comprehensively judge that the simple laboratory abnormality is not clinically significant, it is also allowed to enter the group);
  10. For female subjects of reproductive age, a urine or serum pregnancy test should be performed within 3 days prior to receiving the first study drug administration (day 1 of cycle 1) and the result is negative. If the urine pregnancy test results cannot be confirmed as negative, a blood pregnancy test is requested. Women of non-reproductive age were defined as at least one year after menopause or having undergone surgical sterilization or hysterectomy;
  11. If there is a risk of conception, all subjects (male or female) are required to use contraception with an annual failure rate of less than 1% for the entire duration of treatment up to 120 days after the last study drug administration (or 180 days after the last chemotherapy drug administration).

Exclusion Criteria:

* Other malignant tumors are diagnosed, or oral cancer is not the beginning of neoadjuvant therapy;
* An active autoimmune disease requiring systemic treatment (e.g. use of disease-modifying drugs, glucocorticoids, or immunosuppressants) has occurred within 2 years prior to treatment. Replacement therapies (such as thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic therapy;
* known allogeneic organ transplantation (other than corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
* Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive);
* untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number detected greater than the upper limit of normal value in the laboratory of the study center);

Note: Hepatitis B subjects who meet the following criteria can also be enrolled:

1. HBV viral load <1000 copies /ml (200 IU/ml) before initial dosing, subjects should receive anti-HBV therapy throughout study treatment to avoid viral reactivation;
2. For subjects with anti-HBC (+), HBsAg (-), anti-HBS (-) and HBV viral load (-), prophylactic anti-HBV therapy is not required, but close monitoring of viral reactivation is required;

   * active HCV-infected subjects (HCV antibody positive and HCV-RNA levels above the lower limit of detection);
   * Pregnant or lactating women;
   * The presence of any serious or uncontrolled systemic disease, such as:

1) The resting electrocardiogram has major abnormal rhythm, conduction or morphology, such as complete left bundle branch block, heart block above Ⅱ degree, ventricular arrhythmia or atrial fibrillation; 2) Unstable angina pectoris, congestive heart failure, New York Heart Association (NYHA) grade ≥ 2 chronic heart failure;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2032-08-31 (Estimated)

PRIMARY OUTCOMES:
2 years Event-Free Survival，EFS | 2 years
  2-Year EFS (Event-Free Survival) refers to a key clinical endpoint used in oncology and other medical studies to evaluate the efficacy of treatments. It measures the percentage of patients who remain free of specific negative events for two years after starting treatment. These "events" can include disease progression, recurrence, or treatment-related complications, depending on the study's context.

SECONDARY OUTCOMES:
Overall survival | 5 years
  Overall survival(OS) is the time from day 1 of study treatment(the time randomized) until death from any cause.
Major pathologic response | 6 weeks
  Pathologic response rate to neoadjuvant treatment in resected tumor and lymph nodes. The rate of major pathologic response, defined as <10% residual viable tumor cells in the resection specimen will be compared to historic data with neoadjuvant chemotherapy.
Quality of life assessed by Health-related Quality of Life,HRQoL. | 2 years
  A practical, everyday, functional description of the patient's physical, psychological, and social responses to his or her illness and treatment. This study was evaluated by the Head and Neck Cancer Specific Scale (EORTC QLQ-H&N35)
Objective response rate, ORR | 6 weeks
  Objective tumor response, including CR and PR, was assessed using RECIST version 1.1.
Adverse events rated by NCI-CTCAE v5.0 | 2 years
  The detail number and percentage of adverse events by every systems Assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen memorial hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No